CLINICAL TRIAL: NCT01882348
Title: Changing Pediatric Office Systems Nationally to Address Parental Tobacco Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); American Academy of Pediatrics (Other)
Responsible Party: Principal Investigator, Jonathan P. Winickoff, MD, MPH, Jonathan P. Winickoff, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2013P000777/MGH; R01CA127127 (NIH)
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Tobacco Dependence
Keywords: tobacco control, tobacco treatment, pediatrics, parents
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care Control (No Intervention): Control groups will receive equal number of contacts for training in preparation for enrollment and data collection for the study.
  Clinicians will be given the option to receive a standard American Academy of Pediatrics tobacco control pamphlet to distribute.
  Control groups have the option to receive access to the CEASE online module intervention at the conclusion of the research study which allows practitioners in this group to receive 26 continuing education credit hours.
- Intervention (Experimental): The Intervention Group will receive the CEASE Intervention
  Interventions: Behavioral: CEASE Intervention

INTERVENTIONS:
Behavioral: CEASE Intervention — The CEASE intervention works within existing systems of care to address parental smoking. Elements include (1) Identification of smokers and self-assessment of quitting preferences; (2) Counseling (brief motivational messaging elements include collaborative goal setting, set quit date, personal barriers to quitting, problem-solving strategies, implementing smoke-free homes and cars, and social support, strategies shown to increase satisfaction with the pediatric visit. (3) Medication (NRT prescription and free 1 week supply (while supplies last)-including for those cutting down to quit as recommended in latest guidelines); (4) Quitline enrollment; and (5) Review of CEASE action sheets at each visit until the family is smoke-free.
  Arms: Intervention

SUMMARY:
The proposed study is a Cluster Randomized Controlled Trial designed to test the sustainability of a previously developed, tested, effectively implemented tobacco control strategy-the CEASE intervention, employing state of the art tobacco dependence treatment for parents who smoke.

DETAILED DESCRIPTION:
The CEASE intervention works within existing systems of care to address parental smoking. Based on national guidelines and extensive qualitative research obtained in pilot testing, elements of CEASE can be tailored to work with particular practices' staffing, resources, and physical configuration. CEASE integrates evidence-based tobacco-use screening, cessation assistance, and referral to outside services into visits with families in pediatric clinics. Elements include (1) Identification of smokers and self-assessment of quitting preferences; (2) Counseling (brief motivational messaging elements include collaborative goal setting, set quit date, personal barriers to quitting, problem-solving strategies, implementing smoke-free homes and cars, and social support, strategies shown to increase satisfaction with the pediatric visit.(3) Medication (NRT prescription and free 1 week supply (while supplies last)-including for those cutting down to quit as recommended in latest guidelines); (4) Quitline enrollment via faxed enrollment form; and (5) Review of CEASE action sheets at each visit until the family is smoke-free. We train practices in the adoption, implementation, and maintenance of the intervention. A more detailed training manual discusses additional in-depth strategies for maximizing billing and reimbursement, materials for seasonal cessation opportunities and supporting employees' own cessation efforts.

ELIGIBILITY:
Inclusion Criteria:

* Parents or guardians who smoke or who are former smokers (quit in the last 2 years), are present at the visit, and whose child (any age) is seen by a pediatrician in a participating practice.
* "Smoker" will be defined as answering "yes" to the screening question: "Have you smoked a single cigarette, even a puff, in the past 7 days?"
* "Former smoker" will be defined as answering "no" to the screening question: "Have you smoked a single cigarette, even a puff, in the past 7 days?" and "yes" to the screening question: "Have you quit smoking in the last 2 years?"

Exclusion Criteria:

* Parents under age 18
* Parents who have a child with a medical emergency (any condition requiring transfer for immediate medical intervention)
* Non-consenting individuals
* Non-English speakers
* Prior enrollment in the study during a previous healthcare visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3888 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Delivery of Assistance | over 2 years
  • Delivery of cessation assistance, defined as prescribing medication, or enrolling in the quitline or other program

SECONDARY OUTCOMES:
Change in practice prevalence of parents who smoke | over 2 years
  Change in practice prevalence of parents who smoke assessed at baseline and at 2 years
Parental quit rate | over 2 years
  Change in parental quit rate at the practice: quit in the last 2 years, cotinine-confirmed at baseline and at 2 years
Smokefree homes and cars | over 2 years
  • Reduced parental smoking inside homes and cars assessed by previously validated, self-reported strictly enforced rules prohibiting smoking in the home and car
Parental use of pharmacotherapy or services | over 2 years
  Use of services from any smoking cessation program and/or pharmacotherapy to help quit smoking

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Winickoff, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Nabi-Burza E, Winickoff JP, Drehmer JE, Zeegers MP, Walters BH. A Qualitative Study of Factors Influencing Implementation of Tobacco Control in Pediatric Practices. J Smok Cessat. 2022 May 5;2022:4156982. doi: 10.1155/2022/4156982. eCollection 2022. PMID 35603037
- [Derived] Nabi-Burza E, Drehmer JE, Walters BH, Willemsen MC, Zeegers MPA, Winickoff JP. Smoking Cessation Treatment for Parents Who Dual Use E-Cigarettes and Traditional Cigarettes. J Smok Cessat. 2021 Mar 17;2021:6639731. doi: 10.1155/2021/6639731. eCollection 2021. PMID 34306227
- [Derived] Nabi-Burza E, Wasserman R, Drehmer JE, Walters BH, Luo M, Ossip D, Winickoff JP. Spontaneous Smoking Cessation in Parents. J Smok Cessat. 2021 May 17;2021:5526715. doi: 10.1155/2021/5526715. eCollection 2021. PMID 34306222
- [Derived] Nabi-Burza E, Drehmer JE, Hipple Walters B, Rigotti NA, Ossip DJ, Levy DE, Klein JD, Regan S, Gorzkowski JA, Winickoff JP. Treating Parents for Tobacco Use in the Pediatric Setting: The Clinical Effort Against Secondhand Smoke Exposure Cluster Randomized Clinical Trial. JAMA Pediatr. 2019 Oct 1;173(10):931-939. doi: 10.1001/jamapediatrics.2019.2639. PMID 31403675
- [Derived] Nabi-Burza E, Winickoff JP, Drehmer JE, Gorzkowski JA, Klein JD, Levy DE, Ossip DJ, Regan S, Rigotti NA, Hipple Walters B. Innovations in parental smoking cessation assistance delivered in the child healthcare setting. Transl Behav Med. 2020 Oct 8;10(4):1039-1052. doi: 10.1093/tbm/ibz070. PMID 31157864
- [Derived] Nabi-Burza E, Regan S, Walters BH, Drehmer JE, Rigotti NA, Ossip DJ, Gorzkowski JA, Levy DE, Winickoff JP. Parental Dual Use of e-Cigarettes and Traditional Cigarettes. Acad Pediatr. 2019 Sep-Oct;19(7):842-848. doi: 10.1016/j.acap.2019.04.001. Epub 2019 Apr 11. PMID 30981026
- [Derived] Drehmer JE, Nabi-Burza E, Hipple Walters B, Ossip DJ, Levy DE, Rigotti NA, Klein JD, Winickoff JP. Parental Smoking and E-cigarette Use in Homes and Cars. Pediatrics. 2019 Apr;143(4):e20183249. doi: 10.1542/peds.2018-3249. Epub 2019 Mar 11. PMID 30858346
- [Derived] Drehmer JE, Ossip DJ, Nabi-Burza E, Hipple Walters B, Gorzkowski JA, Winickoff JP. Pediatric Office Delivery of Smoking Cessation Assistance for Breast-Feeding Mothers. Nicotine Tob Res. 2020 Mar 16;22(3):346-353. doi: 10.1093/ntr/nty247. PMID 30521040